CLINICAL TRIAL: NCT07194187
Title: High Intensity Focused Ultrasound (HIFU) Ablation for Treatment of Prostate Tissue in Bladder Outlet Obstruction
Acronym: HIFU for BOO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Michael Palese, Professor, Site Chair Department of Urology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY-24-00513
Record Dates: First submitted 2025-09-09; First posted 2025-09-26 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Bladder Outlet Obstruction; BPH
Keywords: High-intensity focused ultrasound; Interventional; Single Arm; benign prostatic hyperplasia treatment; International Prostate Symptom Score; Device Safety
MeSH Terms: conditions — Urinary Bladder Neck Obstruction

STUDY DESIGN:
Intervention Model Description: This is a single-arm study evaluating the efficacy and safety of the device. All participants will be treated at the same center and will receive the same intervention and follow-up protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Participants with benign prostatic hyperplasia (Experimental): HIFU therapy for benign prostatic tissue ablation in patients with lower urinary tract symptoms (LUTS) due to bladder outlet obstruction
  Interventions: Device: High Intensity Focused Ultrasound

INTERVENTIONS:
Device: High Intensity Focused Ultrasound — High Intensity Focused Ultrasound (HIFU) works with an image-guided transrectal probe that utilizes 3-10 MHz ultrasound waves at very high powers (200W). These waves can be very precisely directed at target tissue. Through both thermal and mechanical forces (shearing motion and mechanical energy leading to hyperthermia) the focal point core temperature can be raised significantly (> 80°C) leading to coagulative necrosis to the target tissue while sparing surrounding tissue. The degree of tissue injury is based on the temperature and the duration of exposure, with the cooling off time allowing for the heat to dissipate to prevent the damage to surrounding tissues. The most common device involves a transrectal transducer with ultrasound guidance that can be performed under either general or spinal anesthesia. The device has been FDA approved to be used in ablation of prostatic tissue since 2018.
  Other Names: HIFU

SUMMARY:
Objectives: To assess the efficacy of HIFU therapy for benign prostatic tissue ablation in patients with lower urinary tract symptoms (LUTS) due to bladder outlet obstruction (BOO) that caused by Benign prostatic hyperplasia (BPH).

The primary objective of the study is to determine the efficacy of HIFU therapy by assessing the changes in IPSS score in 6-month post HIFU procedure for BPH with compared to baseline.

The secondary objectives of this study are as follow:

* To assess any adverse events related to the procedure or device.
* To assess the operation related characteristics including: total operation time and ablation time required in HIFU procedure for BPH, total catheterization time after the HIFU procedure for BPH, and categorical ablation zone
* To assess the patient's post operative pain level at different post op time points.
* To assess the urinary flow and symptoms improvement by studying the changes in IPSS, Qmax, and PVR at different post op time points compared to the baseline.
* To assess the effectiveness of HIFU by studying the changes in PSA levels, types of medication for BPH or any urologic condition, proportion of patients who are taking BPH medication, prostate volume, and prostate calcification level and the reoperation rate within 12-month post-op.
* To assess changes in patients' sexual function at different post op time points.

The hypothesis is that a HIFU ablation is a safe and effective treatment for patients with LUTS due to BOO from BPH.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 45 - 80 diagnosed with LUTS due to BOO from BPH.
* Prostate size > 30cc and < 80cc as measured by transrectal ultrasound (TRUS) or MRI within 1 year prior to treatment.
* A documented history of refusal to take medical therapy, inadequate or failed response to medical therapy, or contraindications to medical therapy.
* Initial baseline International Prostate Symptom Score (IPSS) greater than or equal to 12 which denotes moderate to severe symptoms.
* Baseline peak urinary flow rate (Qmax) of less than 15 mL/s1
* Baseline serum creatinine < 2 mg/dL within 30 days prior to surgery
* Mental capacity, willingness, and ability to sign a study specific informed consent form

Exclusion Criteria :

* BMI > 42
* Patients with an obstructing prostatic median lobe as measured by baseline preliminary imaging and/or confirmed on cystoscopy examination.
* Patients with latex allergies which would permit latex catheterization perioperatively as silicone catheterization is not recommended during HIFU treatment.
* Patients with extensive calcification in the treatment area of the prostate as measured by preoperative imaging with TRUS or MRI and as evaluated by hospital radiology or the principal investigator. Extensive calcification is defined as where the calcification in posterior peripheral zone, which may interfere with experimental treatment procedure, and it is determined by hospital radiologist and further assessed by the PI.
* Patient unable to stop anticoagulants, antiplatelet agents, or NSAIDS (including aspirin > 100mg) prior to treatment which is standard of care.
* Patients using immunosuppressants including corticosteroids (except inhalants) who are unable to withhold medications prior to treatment which is standard of care.
* Known and documented coagulopathy or platelet disorder
* Contraindication to both general and spinal anesthesia which are standard of care.
* Severe illness that would prevent complete study participation.
* History of active or prior treatments for current/suspected PCa.
* Diagnosis of polyneuropathy
* Bladder calculi or bladder diverticulum (pouch size > 20% of full bladder size)
* Active infection, including urinary tract infection or prostatitis.
* Evidence of hydronephrosis on imaging.
* Pre-op urinary catheter uses daily.
* Previous urinary tract surgeries such as, but not limited to prior surgery for LUTS, urinary diversion, artificial urinary sphincter, or penile prosthesis.
* Diagnosis of clinically significant urethral stricture, meatal stenosis, severe phimosis, or bladder neck contracture
* Known damage to the external urinary sphincter.
* Open heart surgery or cardiac arrest < 180 days prior to the date of informed consent
* Known illicit substance abuse.
* Use of anticholinergics (specifically for bladder problems). Use of general anticholinergics is allowed if they do not have documented adverse urinary side effects.
* Dementia or psychiatric conditions which prevent them from completing the required follow up.
* Prior pelvic radiotherapy
* Participation in another ongoing investigational study that could affect responses.
* Unwillingness to accept a transfusion should it be required.
* No members of vulnerable populations will be included in our study.
* History or current diagnosis of chronic prostatitis.
* Diagnosis or prior treatment for chronic pelvic pain syndrome.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-09-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Change in The International Prostate Symptom Score (I-PSS) | baseline and 6 months post-treatment
  The International Prostate Symptom Score (I-PSS) is designed to assess severity of symptoms in benign prostatic hypertrophy. It is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 with higher score indicating more symptomatic. It classifies patients' symptomatology as follows: Mild (symptom score ≤ 7), Moderate (score 8-19), and Severe (score 20-35).

SECONDARY OUTCOMES:
Frequency and proportions of adverse events and all cause hospitalization | within the first 30 days after the HIFU intervention
  Adverse events, probably, or possibly related to the device or surgical procedure, including any all-cause hospitalization within 30 days post-op. Frequencies and proportions of adverse events will be reported in patients likely and unlikely related to the device or surgical procedure.
Operation time | approximately 45-120 minutes
  Operation time: Amount of time required from the start to the end of the HIFU procedure, the total operation time
Ablation time | average 15-45 minutes
  Ablation time: Amount of time required for HIFU to ablate the benign prostatic tissue. Defined as the time from the first HIFU firing until the time of the last HIFU firing.
Catheterization times | 1 week post-procedure, or until the patient passes the trial of void
  Catheterization times: Number of days required for foley catheter after the procedure.
Categorical Ablation Zones (Peripheral, Transitional, or Central Prostate Zones) | During procedure
  Categorical ablation zones: Defined as the prostate area involved in HIFU ablation, including the peripheral, transitional, or central zone. This outcome will be recorded as a categorical variable based on the anatomical region(s) of the prostate targeted by the ablation.
Male-Genitourinary Pain Index (M-GUPI) pain questionnaire | at discharge after HIFU procedure (expected time: Post-op Day 1), 1-week and 1-month post-op
  Patient's post-op pain level will be assessed using the M-GUPI pain questionnaire: a pain questionnaire to assess their postoperative pain. Total score of the M-GUPI will be analyzed along with patients' use of opioid pain medication to assess patient pain levels at discharge after HIFU procedure.
  The M-GUPI questionnaire has 10 pain items (total pain subscale score 0-23), 2 urinary symptom items (total urinary subscale score 0-10), and 3 QOL items (total QOL subscale score 0-12). As with the NIH-CPSI, the scores from each item are summed for a total score that ranges from 0 to 45, higher scores indicate greater severity.
Changes in IPSS scores | Baseline, 1-, 3-, 12- months post-treatment
  Symptoms and urinary flow improvement are assessed through changes in IPSS scores: Difference in IPSS scores at 1 month, 3 months, and 12 months post-treatment compared to pre-op baseline. IPSS score is a standardized questionnaire for assessing urinary flow. The total score can range from 0 to 35 (asymptomatic to very symptomatic). It classifies patients' symptomatology as follows: Mild (symptom score ≤ 7), Moderate (score 8-19), and Severe (score 20-35).
Changes in maximum flow rate (Qmax) | Baseline, 1-, 3-, 6-, 12- months post-treatment
  Symptoms and urinary flow improvement are assessed through changes in Qmax .
  Qmax is the maximum flow rate of urine, measured in milliliters per second (ml/s). A Qmax value below 15 ml/s may suggest urinary issues
Changes in Post-Void Residual (PVR) | Baseline, 1-, 3-, 6-, 12- months post-treatment
  Symptoms and urinary flow improvement are assessed through changes in PVR. PVR is the amount of urine left in the bladder after urination.
Changes in the type of BPH medications | Baseline, 1 week, 1-, 3-, 6-, and 12- month post-treatment
  Effectiveness of HIFU is assessed through changes in the type of BPH medications and proportions of patients who are taking BPH medications following treatment compared to pre-op baseline BPH medications at discharge after HIFU procedure, 1 week, 1-, 3-, 6-, and 12- month post op follow up. Types of BPH medications include Flomax, Uroxatral, Cardura, Rapaflo, Hytrin, Proscar, Propecia, Avodart.
Change in Prostate Specific Antigen (PSA) level. | Baseline, 6-, and 12- month post-treatment
  Effectiveness of HIFU is assessed through change from pre-op baseline PSA to PSA at 6-month and 12-month post op.
  Prostate-specific antigen (PSA) is a protein produced by prostate cells. The PSA test is done to help screen for and monitor prostate cancer in men.
Change in Prostate measurement | Baseline, 6-, and 12- month post-treatment
  Effectiveness of HIFU is assessed through change from pre-op baseline prostate measurement to 6- to 12- month post-op. Pre-op baseline measurement will be defined as within 1 year prior to the HIFU BPH procedure. This will be performed through transrectal ultrasound or MRI scan to measure the size of prostate gland and assess the calcification level of prostate. If patients have both imaging results, MRI values will be favored for more accurate assessment. Post operative imaging will be assessed in between 6 to 12 months post-op and compared with the pre-op baseline imaging result. Differences of the prostate size and calcification level between 6-12 months post-op versus pre-op baseline will be collected.
Number of BPH procedures | 12- month post-treatment
  Effectiveness of HIFU is assessed through re-operation rate at 12 months: number of BPH procedures that patient required after the HIFU procedure.
Change in the International Index of Erectile Function (IIEF) questionnaire | Baseline, 3- and 6- months post treatment
  Difference in erectile or ejaculation dysfunction in patients who are sexually active in baseline pre-op:
  Difference in IIEF score at 3-months post-op minus pre-op baseline and at 6-month post-op minus pre-op baseline. The International Index of Erectile Function is a validated questionnaire used to assess patients' erectile function and is standard of care to assess prior to and following BOO treatment to measure treatment success and complications. Erectile dysfunction severity is classified as follows based on the score: 1-10 indicates severe dysfunction; 11-16, moderate dysfunction; 17-21, mild to moderate dysfunction; 22-25, mild dysfunction; and 26-30, no dysfunction. Total score ranges from 15-75, total score indicates better health outcomes.
Change in the Male Sexual Health Questionnaire- Ejaculatory Dysfunction (MSHQ-EjD) | Baseline, 3- and 6- months post treatment
  Difference in erectile or ejaculation dysfunction in patients who are sexually active in baseline pre-op: Difference in MSHQ-EjD scores at 3-months post-op minus baseline and at 6-month post-op minus pre-op baseline. The Male Sexual Health Questionnaire- Ejaculatory Dysfunction is a validated questionnaire used to assess patients' ejaculatory function and is standard of care to assess prior to and following BOO treatment to measure treatment success and complications. Scores range from 0 to 20, higher scores indicate better health outcomes. Scores below 8 suggest potential ejaculatory dysfunction, including premature or delayed ejaculation. Scores between 9 and 12 indicate moderate concerns that may not meet clinical criteria for dysfunction. Scores above 12 generally reflect normal ejaculatory function with minimal concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Palese, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Union Square, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. For individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link tbd).